CLINICAL TRIAL: NCT05318209
Title: Comparison Between Closed-chain Shoulder Girdle Scapular Depression Exercise and Shoulder Girdle Depression Against Manual Resistance on Patients With Shoulder Impingement Syndrome
Brief Title: Effect of Closed-chain Shoulder Girdle Scapular Depression Exercise on Shoulder Impingement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nasr Awad Abdelkader Othman (Other)
Collaborators: Atef Abdulalim Nadier, Pharos University (Unknown); Ehab Ai Abdalah,Lecurer, Horus University (Unknown)
Responsible Party: Sponsor-Investigator, Nasr Awad Abdelkader Othman, Assistant Professor,Department of Physical Therapy for Musculoskeletal Disorders, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/003377
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study grou[p (Experimental): Closed-chain shoulder girdle scapular depression exercise
  Interventions: Other: Exercise
- control group (Active Comparator): Shoulder girdle depression against manual resistance exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Closed-chain Shoulder Girdle Scapular Depression Exercise

SUMMARY:
forty patients will be assigned randomly into 2 equal groups Study group (n=23) will receive "closed-chain shoulder girdle scapular depression exercise" in addition to Stretching for posterior capsule & pectoralis minor, Eccentric exercise for external rotators and Strength exercises for serrates anterior and low intensity ultrasound Control group B (n=23) will receive "shoulder girdle depression against manual resistance exercise" in addition to stretching for posterior capsule & pectoralis minor, eccentric exercise for external rotators and Strength exercises for serrates anterior and low intensity ultrasound .

The exercise program will consist of 3 sessions / week for 5 weeks

DETAILED DESCRIPTION:
BACKGROUND:

Patients with shoulder impingment syndrome report disability, especially during overhead movements, which may hinder activities of daily living .

Muscular strengthening training influences the resting position and scapular movement pattern of subjects with shoulder impingement syndrome and improve function of the affected shoulder.

Therefore, the focus of treatment for the syndrome is on performing exercises, including stretching, strengthening, and neuromuscular control exercises.

Although multiple types of exercise, such as scapular stability exercises, strengthening of the rotator cuff through range, and flexibility exercises for the anterior and posterior shoulder exercise is effective in the management of patients with shoulder impingement syndrome, there is not enough evidence to say whether one mode of exercise is superior to another.

RESEARCH QUESTION:

Are there any difference between closed-chain shoulder girdle scapular depression exercise and shoulder girdle depression against manual resistance exercise on patients with shoulder impingement syndrome

METHODS:

forty patients will be assigned randomly into 2 equal groups Study group (n=23) will receive "closed-chain shoulder girdle scapular depression exercise" in addition to Stretching for posterior capsule & pectoralis minor, Eccentric exercise for external rotators and Strength exercises for serrates anterior and low intensity ultrasound Control group B (n=23) will receive "shoulder girdle depression against manual resistance exercise" in addition to stretching for posterior capsule & pectoralis minor, eccentric exercise for external rotators and Strength exercises for serrates anterior and low intensity ultrasound .

The exercise program will consist of 3 sessions / week for 5 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 25 to 45 years old.
* Patients with shoulder impingement stage I &II as judged by criteria of neer classification.
* Patients diagnosed by orthopedic surgeon with shoulder impingement, the diagnosis will be confirmed by positive Neer and Hawkins tests.

Exclusion Criteria:

* History of cardiac diseases or dyspnea on exertion
* Patients with cervical radiculopathy.
* Patients with shoulder instability.
* Patients with frozen shoulder.
* Acute shoulder trauma.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain will be measured by visual analogue scale | 10 minutes
  10cm visual analogue scale (0= no pain, and 10= maximum pain) will be used to determine overall shoulder pain

SECONDARY OUTCOMES:
Range of motion (flexion and abduction) will be measured by Electronic goniometer | 20 minutes
  Electronic Goniometer will be used to measure shoulder range of motion (Flexion and abduction)
Function | 30 minutes
  shoulder function will be measured by western Ontario Rotator Cuff Questionnaire (WORC).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr Elshiekh Hospital, Kafr ash Shaykh, Egypt